CLINICAL TRIAL: NCT03232736
Title: Randomized interventiOn of Biventricular Pacemaker Function on ventrIcular Function Among Patients With mechaNical Circulatory Support Devices
Brief Title: InterventiOn of Biventricular Pacemaker Function on ventrIcular Function Among Patients With LVAD's
Acronym: ROBIN
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1042
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Heart Diseases; Left Ventricular Dysfunction
MeSH Terms: conditions — Heart Diseases; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Individuals free of cardiovascular disease and not on any medications to treat a cardiovascular-related condition
- LVAD Group: Individuals with history of advanced heart failure who are supported by left ventricular assist devices

SUMMARY:
The primary reason the investigators are doing this study are to understand how the right side of the heart functions in heart failure patients with left ventricular assist devices (LVADs, or "mechanical hearts"). Second, the investigators are interested in understanding how different pacemaker settings influence function of the heart at rest and activity.

DETAILED DESCRIPTION:
Healthy individuals, as well as patients with advanced heart failure supported by LVADs, completed invasive hemodynamic analysis at rest and with exercise to characterize right-sided heart function at rest and with exercise during invasive cardiopulmonary exercise testing on upright cycle ergometry.

ELIGIBILITY:
15 patients with advanced heart failure (HF) who have already undergone implantation of a continuous-flow left ventricular assist device (CF-LVAD) implantation.

Inclusion criteria:

1. Have already received CF-LVADs and are clinically stable,
2. Ambulatory outpatients and are fully recovered (at least 3 months) from LVAD implantation;

Exclusion criteria:

1. Individuals with clinical right ventricular (RV) failure under resting conditions, defined as moderate-severely reduced RV systolic function on echocardiography, or
2. Clinical evidence of RV failure (elevated jugular venous pressures, 3 or 4+ [significant] peripheral edema);
3. Disorders that adversely influence exercise ability (e.g. arthritis, peripheral vascular disease, pulmonary disease); and

10 healthy individuals will serve as a control group to define normal RV function during exercise.

Inclusion criteria:

1) Persons without a past medical history of cardiovascular disease or related disease such as:

1. hypertension,
2. diabetes,
3. peripheral vascular disease,
4. arrhythmias,

f. are not taking any cardiac-related medications (e.g. antihypertensive medications).

Exclusion criteria:

1. Individuals requiring systemic anticoagulation with vitamin-K antagonists or new/direct oral anticoagulants ("NOAC"/"DOAC");
2. Disorders that adversely influence exercise ability (e.g. arthritis, peripheral vascular disease).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 patients with advanced HF who have already undergone CF-LVAD implantation.
  10 healthy individuals will serve as a control group to define normal RV function during exercise.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Cornwell, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornwell WK, Tran T, Cerbin L, Coe G, Muralidhar A, Hunter K, Altman N, Ambardekar AV, Tompkins C, Zipse M, Schulte M, O'Gean K, Ostertag M, Hoffman J, Pal JD, Lawley JS, Levine BD, Wolfel E, Kohrt WM, Buttrick P. New insights into resting and exertional right ventricular performance in the healthy heart through real-time pressure-volume analysis. J Physiol. 2020 Jul;598(13):2575-2587. doi: 10.1113/JP279759. Epub 2020 May 18. PMID 32347547
- [Background] Tran T, Muralidhar A, Hunter K, Buchanan C, Coe G, Hieda M, Tompkins C, Zipse M, Spotts MJ, Laing SG, Fosmark K, Hoffman J, Ambardekar AV, Wolfel EE, Lawley J, Levine B, Kohrt WM, Pal J, Cornwell WK 3rd. Right ventricular function and cardiopulmonary performance among patients with heart failure supported by durable mechanical circulatory support devices. J Heart Lung Transplant. 2021 Feb;40(2):128-137. doi: 10.1016/j.healun.2020.11.009. Epub 2020 Nov 22. PMID 33281029

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control: healthy individuals free of cardiovascular disease and not on any cardiac-related medications, age > 18years.
- LVAD Group w/Pacemaker: Pacemaker adjustments will be made to this group in blinded manner.
  Pacemaker adjustments: LVAD subjects with CRT device will have leads turned both on and off in blinded manner
  CRT: CRT device
Period: Overall Study
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Started | 9 | 13
Completed | 9 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy individuals are those who are free of cardiovascular disease and not on any medications to treat a cardiovascular disease. Patients with LVADs are those with a history of advanced heart failure who are supported by an LVAD
Groups:
- Healthy Control: Healthy controls free of heart disease and not on any medications. Age 18+ years
- LVAD Group: Heart failure patients supported by LVAD
- Total: Total of all reporting groups
Arm/Group | Healthy Control | LVAD Group | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 61 (9) | 52 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 12 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 13 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Peak Vo2
Description: peak Vo2 measured by indirect calorimetry during cardiopulmonary exercise testing
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Healthy Control: healthy people free of heart disease.
- LVAD Group w/Pacemaker: heart failure patients supported by an LVD.
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
ml/kg/min | 33 (10.4) | 12.5 (3.2)

2. Primary Outcome: Cardiac Output
Description: cardiac output measured during invasive cardiopulmonary exercise testing.
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Healthy Control: healthy people without cardiac disease
- LVAD Group w/Pacemaker: heart failure patient supported by lvads.
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
L/min | 18.4 (7.3) | 9.1 (3.3)

3. Secondary Outcome: Blood Pressure
Description: mean arterial pressure during exercise
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Healthy Control | LVAD Group
Number analyzed (Participants) | 9 | 13
mmHg | 119 (7) | 91 (10)

4. Secondary Outcome: Respiratory Exchange Ratio
Description: Respiratory exchange ratio derived from indirect calorimetry
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
ratio | 1.08 (0.08) | 0.03 (0.08)

5. Secondary Outcome: Minute Ventilation
Description: Minute ventilation during cardiopulmonary exercise testing
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
L/min | 102 (40) | 56 (19)

6. Secondary Outcome: Tau
Description: unit of measure of diastolic function during exercise
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
msec | 25 (6) | 54 (49)

7. Secondary Outcome: Stroke Work
Description: stroke work during exercise
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: mmHg*mL
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
mmHg*mL | 4999 (2342) | 2455 (783)

8. Secondary Outcome: EES/EA
Description: ventricular arterial coupling during exercise
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
Number analyzed (Participants) | 9 | 13
ratio | 1.6 (0.8) | 1.40 (0.34)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Groups:
- LVAD Group w/Pacemaker: Heart failure patients supported by an LVAD.
Arm/Group | Healthy Control | LVAD Group w/Pacemaker
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 0/9 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT03232736/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03232736/ICF_001.pdf